CLINICAL TRIAL: NCT05781048
Title: An Open-label, Multi-center Phase I Study of Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of HRS-6209 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Phase I Clinical Study of the Safety， Tolerability，Pharmacokinetics, and Initial Efficacy of HRS-6209 Monotherapy in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6209-I-101
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-6209 (Experimental)
  Interventions: Drug: HRS-6209

INTERVENTIONS:
Drug: HRS-6209 — HRS-6209

SUMMARY:
The study is being conducted to evaluate the efficacy, andsafety of HRS-6209in subjects with advanced solid tumors.To explore the reasonable dosage of HRS-6209.This study also preliminarily evaluated the efficacy of HRS-6209 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing to participate in the study, sign the informed consent form, have good compliance, and cooperate with follow-up visits.
2. Aged 18-80 years, male or female
3. Patients with advanced malignant tumors confirmed pathologically;
4. Failure of adequate standard treatment, or no effective standard treatment;
5. Patients must have at least 1 extracranial measurable target lesion per RECIST v1.1 ;
6. The expected survival period is more than 12 weeks;
7. The Eastern Cooperative Oncology Group (ECOG) physical fitness score is 0 - 1;
8. Have sufficient bone marrow and organ function (have not received blood transfusion or hematopoietic stimulating factor treatment within 14 days)；
9. Female subjects of childbearing age must undergo a serum pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraception during the study period and within 6 months after the last administration of the study drug Measures: For male subjects whose partners are females of childbearing age, they should be surgically sterilized, or agree to use effective methods of contraception during the study period and within 3 months after the last study administration;

Exclusion Criteria:

1. Subjects with a history of malignant tumors, except patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or cervical carcinoma in situ who have undergone possible curative treatment and did not have disease recurrence within 3 years since starting the treatment；
2. Subjects had cancerous meningitis or untreated central nervous system metastases
3. Subjects experienced intestinal obstruction and gastrointestinal perforation within 3 months prior to initial medication
4. There is third-space effusion that cannot be controlled by drainage and other methods (such as massive ascites, pleural effusion, pericardial effusion)；
5. Subjects had clinical cardiac symptoms or disease that was not well controlled within 6 months prior to initial medication
6. Subjects had or currently had idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia , drug pneumonia, or CT during screening showed active pneumonia；
7. Arteriovenous thrombosis occurred within 6 months prior to the first dose
8. Severe infection occurred within 4 weeks prior to initial administration
9. During the screening period/before the first administration, fever of unknown origin> 38.5°C
10. Known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS)
11. Subjects had active hepatitis；
12. Subjects received live attenuated vaccine within 4 weeks or planned for the study period prior to initial administration；
13. Subjects were scheduled to receive other systemic antitumor therapies during the study period；
14. Participated in other clinical studies within 4 weeks before starting the study drug treatment；
15. Subjects were unable to swallow pills or capsules normally, or had gastrointestinal abnormalities that the researchers determined might affect drug absorption；
16. Other factors as judged by the investigator that may lead to the termination of the study, such as other serious diseases, serious laboratory test abnormalities, or family or social factors that could affect the safety of the subject, or the collection of study data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: Number of subjects with adverse events and the severity of adverse events | every 4 weeks after treatment initiation，up to approximately 2 years.
DLT(Dose-limiting toxicity） | during the first 30-day cycle of SHR-6209 treatment
MTD（Maximum tolerated dose） | 4 weeks after treatment initiation
RP2D（Recommended Phase II Dose） | 4 weeks after treatment initiation

SECONDARY OUTCOMES:
ORR（Objective response rate (ORR) - RECIST 1.1 | Up to approximately 6 months
  ORR is defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR) according to RECIST 1.1）
DoR（Duration of Response (DoR)Duration of Response (DoR) per RECIST 1.1） | Up to approximately 2 years
DCR（Disease control rate（DCR）-RECIST 1.1 | Up to approximately 2 years
  DCR is defined as the proportion of subjects who have achieved Stable disease(SD)、complete response (CR) or partial response (PR) according to RECIST 1.1）
PFS-Progression-free survival(PFS) PFS per RECIST 1.1 | Up to approximately 2 years

IPD SHARING:
Plan to Share IPD: Undecided